CLINICAL TRIAL: NCT01990508
Title: Randomized Trial of Financial Incentives to Reduce Sugar-sweetened Beverage Purchases by Low-income, Latino Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Anne N. Thorndike, MD, MPH, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2013P001130
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Obesity Prevention
Keywords: sugar-sweetened beverages; traffic-light labels; financial incentives; low-income community; obesity prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Targeted beverage education and financial incentives (Experimental): Study subjects receive monthly letters with beverage education and financial incentives for not purchasing sugar-sweetened beverages
  Interventions: Behavioral: Targeted beverage education and financial incentives; Behavioral: Traffic-light labeling of all beverages in store
- Control (Sham Comparator): Monthly letters with generic nutrition information only
  Interventions: Behavioral: Traffic-light labeling of all beverages in store

INTERVENTIONS:
Behavioral: Targeted beverage education and financial incentives
  Arms: Targeted beverage education and financial incentives
Behavioral: Traffic-light labeling of all beverages in store — All beverages in the supermarket will be labeled as red, yellow, or green

SUMMARY:
Approximately 15% of the US population is enrolled in the Supplemental Nutrition Assistance Program (SNAP), and 50% are children. Although the goal is to improve nutritional health, preliminary data suggest that enrollment in SNAP is associated with obesity and metabolic risks and that SNAP reimburses $4 billion annually for sugar-sweetened beverages (SSBs). This pilot project tests an innovative strategy to reduce purchase of non-nutritive, SSBs by low-income families with children by combining targeted point-of-purchase education with a randomized trial of financial incentives to discourage purchase of unhealthy beverages. The study will take place at a mid-size grocery store that is located in a low-income, Latino community and where 30% of purchases are made with SNAP. Targeted beverage education will be provided to all study subjects with a traffic-light system to identify healthy and unhealthy beverages at the point-of-purchase. Individual beverage purchases will be tracked by electronically stored cash register sales. Supplementary validation of beverage consumption will be assessed by 24 hour dietary recall. Aim 1 is to conduct a randomized controlled trial to compare purchase and consumption of SSBs by families assigned to a financial incentive to reduce purchase of SSBs with families assigned to control (no incentives). Aim 2 is to compare the purchase of SSBs by families in both arms during the study period when they are exposed to the traffic-light system to a baseline period prior to traffic-light education. Results of this project will provide pilot data for larger scale interventions to promote healthy choices among low-income families.

ELIGIBILITY:
Inclusion Criteria:

* purchase >75% of groceries at targeted supermarket (regular customer)
* at least one child <= 18 years old living at home

Exclusion Criteria:

* not fluent in Spanish or English
* no address or phone for contact

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Purchase of sugar-sweetened beverages | 4 months

SECONDARY OUTCOMES:
Consumption of sugar-sweetened beverages | 4 months

OTHER OUTCOMES:
Purchase of red-labeled beverages | 6 months
  Pre-post evaluation of purchase of red-labeled beverages before and after the labels are in place

CONTACTS AND LOCATIONS:
Overall Officials: Anne N Thorndike, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Franckle RL, Levy DE, Macias-Navarro L, Rimm EB, Thorndike AN. Traffic-light labels and financial incentives to reduce sugar-sweetened beverage purchases by low-income Latino families: a randomized controlled trial. Public Health Nutr. 2018 Jun;21(8):1426-1434. doi: 10.1017/S1368980018000319. Epub 2018 Mar 1. PMID 29493476